CLINICAL TRIAL: NCT05716152
Title: Assessment of Serum Testosterone and Tissue Androgen Receptors in Male Patients With Psoriasis Vulgaris
Brief Title: Hormonal Associations in Male Patients With Psoriasis Vulgaris
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelhamed Mohamed, Principal Investigator & resident of dermatology in sohag general hospital,, Sohag University
Other Study IDs: Soh-Med-22-11-07
Record Dates: First submitted 2023-01-14; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Psoriasis vulgaris participants
  Interventions: Diagnostic Test: Morning blood sample and skin punch biopsy of 4 mm diameter.
- not diseased participants
  Interventions: Diagnostic Test: Morning blood sample and skin punch biopsy of 4 mm diameter.

INTERVENTIONS:
Diagnostic Test: Morning blood sample and skin punch biopsy of 4 mm diameter. — 1. Morning blood sample (8:00-10:00 am) will be obtained for assessment of Total Testosterone (TT), Free Testosterone (fT), Luteinizing hormone (LH), Follicle stimulating hormone (FSH), and Estradiol (E2).
  2. Skin biopsy:
  Skin punch biopsy of 4 mm diameter will be obtained from both psoriasis patients (from the lesional and non-lesional sites), and the control group (normal skin). Tissue specimens will be used for formation of Paraffin embedded blocks. Slides will be stained by routine Hematoxylin and Eosin stain. The expression of AR will be measured by immune and histochemical staining by the use of a mouse monoclonal antibody

SUMMARY:
A cross sectional clinical study will be conducted on male patients with moderate and sever psoriasis vulgaris to:

* Identify the pattern of serum testosterone level and tissue androgen receptors.
* Evaluate the relationship between serum testosterone level, tissue androgen receptors and the severity of psoriasis vulgaris

DETAILED DESCRIPTION:
A prospective cross sectional clinical study will be conducted on (51) male patients with clinically diagnosed psoriasis vulgaris seeking medical advice at Dermatology outpatient clinics, Sohag University Hospital, Sohag. Age matched healthy adults (51) will be recruited as a control group. The study design will be approved by the ethical and scientific research committee of Sohag University. An informed consent will be obtained from all patients. Dignosis of psoriasis will be confirmed by Dermoscopy.

1. Initial evaluation:

   History taking of patients will include personal history, special habits, and drug treatment. General examination will include weight, height, BMI, and blood pressure.
2. Dermatological evaluation:

   The Psoriasis Area Severity Index (PASI) will be used for patients' evaluation as it is currently the most popular tool in clinical studies. It is a measure of the average redness, thickness and scales of the lesions (each graded on a 0-4 scale), weighed by the area of involvement. The final result of this method of assessment ranges from (0.0 to 72.0). Severity of plaque psoriasis will be graded to mild (PASI ≤10) and moderate to severe (>10). Only patients with moderate to severe plaques psoriasis will be included.
3. Hormonal assessment:

   3-1- Androgen deficiency screening: The Arabic version of the Aging Male Symptoms (AMS) score will be used for Androgen deficiency screening . The AMS questionnaire includes 17 questions which are scored from 1 to 5 for each. It has 3 dimensions, i.e. psychological, somatic, and sexual subscale. The total score is the sum of the three-dimension scores which ranges from 17 to 85. The total AMS score is defined as 'no/little' (17-26 points), 'mild' (27-36 points), 'moderate' (37-49 points), and 'severe' (≥50 points). 3-2- Hormonal laboratory investigations: Morning blood sample (8:00-10:00 am) will be obtained for assessment of Total Testosterone (TT), Free Testosterone (fT), Luteinizing hormone (LH), Follicle stimulating hormone (FSH), and Estradiol (E2).
4. Other laboratory investigations:

   4-1- Lipid profile assessment: Blood sample will be taken after overnight fasting (12-14 hours) to assess triglyceride, total cholesterol, High-density lipoprotein (HDL), and Low-density lipoprotein (LDL). 4-2- C-Reactive protein (CRP): as a marker of chronic inflammation.
5. Skin biopsy:

Skin punch biopsy of 4 mm diameter will be obtained from both psoriasis patients (from the lesional and non-lesional sites), and the control group (normal skin). Tissue specimens will be used for formation of Paraffin embedded blocks. Slides will be stained by routine Hematoxylin and Eosin stain. The expression of AR will be measured by immune and histochemical staining by the use of a mouse monoclonal antibody.

Sample size calculation:

Sample size calculation was carried out using G*Power 3 software. A calculated minimum sample of 102 participants in 1:1 design (51 male patients with psoriasis vulgaris as cases and 51 age matched control) will be needed to detect an effect size of 0.5 in the mean level of total testosterone and AR expression, with an error probability of 0.05 and 80% power on a two-tailed test.

ELIGIBILITY:
Inclusion Criteria:

Cases:

* Male patients with plaque psoriasis.
* With clinically moderate to severe plaque psoriasis (PASI score >10).
* For at least 1 year.
* Age (18-55) years old.

Control:

●Healthy male volunteers matched to the patient group for age and sex.

Exclusion Criteria:

* Other clinical varieties of psoriasis.
* History of diabetes mellitus.
* History of advanced renal or hepatic disease.
* History of genital disorders, or hormonal impalance.
* Current use of hormonal therapy, lipid-reducing drugs, and/or gluco- corticosteroid.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cases:
  ✔Male patients with clinically moderate to severe plaque psoriasis (PASI score >10) for at least 1 year and age (18-55) years old.
  Control:
  ✔Healthy male volunteers matched to the patient group for age and sex.
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Blood sample. | 1.5 year
  Morning blood sample (8:00-10:00 am) will be obtained for assessment of Total Testosterone (TT), Free Testosterone (fT), Luteinizing hormone (LH), Follicle stimulating hormone (FSH), and Estradiol (E2).
Skin biopsy | 1.5 year
  Skin punch biopsy of 4 mm diameter will be obtained from both psoriasis patients (from the lesional and non-lesional sites), and the control group (normal skin). Tissue specimens will be used for formation of Paraffin embedded blocks. Slides will be stained by routine Hematoxylin and Eosin stain. The expression of AR will be measured by immune and histochemical staining by the use of a mouse monoclonal antibody

IPD SHARING:
Plan to Share IPD: Yes